CLINICAL TRIAL: NCT01450553
Title: Research and Development Study: Tissue Collection From Patients Who Are Undergoing Surgery for Non-Small Cell Lung Cancer
Brief Title: Tissue Collection Study for Patients With Non-Small Cell Lung Cancer With Resectable Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Precision Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: RD-110
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Tissue Collection; Lung Cancer; Non-Small Cell Lung Cancer; Early Stage Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human tumor tissues will be collected and preserved in three different tissue formats:
  * Fresh Frozen
  * FFPE
  * RNAlater
Oversight: Data Monitoring Committee: No

SUMMARY:
A 15-gene lung signature was created to identify predictive and prognostic biomarkers for Non-Small Cell Lung Cancer (NSCLC) patients. The 15-gene signature was validated using a microarray platform with fresh frozen tumor tissue to place NSCLC patients into high risk and low risk cohorts with significantly different survivals.

Using fresh frozen tissue can be challenging, so this study attempts simplify the process by migrating the 15-gene signature from fresh frozen to two alternative tissue formats: Formalin Fixed Paraffin Embedded (FFPE) and RNAlater.

The gene expressions of the different tissue formats will be compared to see if the fresh frozen tissue results are similar to the alternative tissue formats.

DETAILED DESCRIPTION:
Patients with early stage NSCLC will be consented prior to surgery so that any excess tissue collected during surgery can be collected in one of the three tissue formats (Fresh Frozen, FFPE, RNAlater) and sent to the Sponsor for testing.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of stage I or II Non-Small Cell Lung Cancer (NSCLC)
* Must have resectable disease and complete surgical resection planned
* Histologically or cytologically confirmed adenocarcinoma, squamous or large cell carcinoma NSCLC
* No prior chemotherapy, biologic/molecular targeted therapy or radiation therapy for this cancer
* Tumor specimen samples must be collected within 1 hour of surgery
* Patient must be at least 18 years of age
* Patient must sign and date an approved study consent form

Exclusion Criteria:

* Patients with psychiatric or addictive disorders that would preclude obtaining study consent
* Informed consent obtained the same day as surgery
* Absence of histological diagnosis of lung cancer
* Known infectious disease
* History of chemotherapy, biologic/molecular targeted therapy or radiation therapy for this cancer or any prior cancer or any other non-cancer diseases or illnesses, i.e. rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-Small Cell Lung Cancer patients undergoing surgery for resection of disease from hospital based locations.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2011-10

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cardio-Thoracic Surgeons, P. C., Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Martin Memorial Treasure Coast Surgeons, Stuart, Florida
  - Baptist Hospital East, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Centennial Thoraic Surgeons, Nashville, Tennessee